CLINICAL TRIAL: NCT06020092
Title: Histological Analysis of Osteogenic Potential of Biphasic Calcium Phosphate in Alveolar Ridge Augmentation
Brief Title: Histological Analysis of Osteogenic Potential of Biphasic Calcium Phosphate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Marija Čandrlić, Postdoctoral researcher at Department of Dental Medicine, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2158-61-46-22-109
Record Dates: First submitted 2023-08-10; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Alveolar Ridge Enlargement; Fenestration; Dehiscence
Keywords: bone regeneration; alloplast; bovine xenograft; guided bone regeneration
MeSH Terms: interventions — benzo(c)phenanthrene-5,6-imine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable biphasic calcium phosphate (maxresorb inject, botiss GmbH) (Experimental): This biomaterial is an alloplastic bone substitute material in the form of a paste that is placed into the defect with a plastic syringe. The material consists of an aqueous gel containing granules of biphasic calcium phosphate in the composition of 60% HA and 40% β-TCP (particle size between 15-50 nm).
  Interventions: Procedure: Bone augmentation with I-BCP
- Bovine xenograft (cerabone, botiss GmbH) (Active Comparator): The material is completely anorganic and consists of 100% HA. For this study, the material will be used in granular form (the size of the granules is between 0.5 and 1 mm), mixed with physiological solution prior to placement into the defect.
  Interventions: Procedure: Bone augmentation with BX

INTERVENTIONS:
Procedure: Bone augmentation with I-BCP — The extraction socket will be filled after tooth extraction with I-BCP, in order to achieve bone regeneration and prevent volume loss after tooth extraction.
  Arms: Injectable biphasic calcium phosphate (maxresorb inject, botiss GmbH)
Procedure: Bone augmentation with BX — The extraction socket will be filled after tooth extraction with BX, in order to achieve bone regeneration and prevent volume loss after tooth extraction.
  Arms: Bovine xenograft (cerabone, botiss GmbH)

SUMMARY:
Bone healing after tooth extraction may be affected by defects in the buccal wall of the alveolus, such as fenestrations and dehiscences. Therefore, it is advisable to perform a surgical procedure such as guided bone regeneration after tooth extractions. Different biomaterials are used for this purpose. The aim of this study is to investigate the qualitative and quantitative histological changes in human biopsies taken after 6 months of healing of extraction sockets with buccal wall defects. For this purpose, the defects of 36 patients (18 per group) will be augmented with injectable biphasic calcium phosphate (I-BCP) or bovine xenograft (BX) after extraction. After six months of healing, bone biopsies will be taken and processed to the qualitative and quantitative histological analysis.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled clinical trial. To participate in the study, patients requires to have at least one tooth predisposed to extraction and to have a dental implant placed after completion of the healing period. The indications for tooth extraction are: chronic periapical process, chronic periodontal disease, or fracture of the vertical bone. The inclusion criteria are: age between 18 and 60 years, intact physical and mental health, patient must understand the study protocol, patient must sign an informed consent. Patients will be excluded from the study if they had at least one of the absolute contraindications to implant prosthetic therapy described by Wang and Hwang. Other exclusion criteria included the following systemic diseases: uncontrolled diabetes, osteoporosis and osteopenia, and vitamin D deficiency, bisphosphonate therapy, glucocorticoid therapy, hypothyroidism, uncontrolled cardiovascular disease (hypertension, coronary artery disease, congestive heart failure), and the following local factors: use of tobacco products (up to 10 cigarettes per day) and poor oral hygiene. Pregnant and lactating women will not included in the study.

In addition to the general health criteria mentioned above, the patient has to meet at least one intraoral criterion, namely the presence of a buccal bone defect such as fenestration or dehiscence. Patients who met the inclusion criteria and were willing to participate, are randomly assigned via a web interface (https://www.randomizer.org/).

Participants and materials Participants will be recruited from the oral surgery office. A total of 36 healthy patients will be included in the study. In analyzing the validity of the test, the approach of equivalence of the tested methods and noninferiority of the tested method compared with the existing method was used. With a significance level α of 0.05, a test power of 80%, an expected standard deviation of the predicted result of 10, and an equivalence limit of d = 10, it was necessary to include at least 36 subjects in the study, 18 subjects per group.

A total of 18 patients in the test group will receive I-BCP (Maxresorb® inject, Botiss GmbH, Berlin, Germany). This biomaterial is an alloplastic bone substitute material in the form of a paste that is placed into the defect with a plastic syringe. The material consists of an aqueous gel containing granules of biphasic calcium phosphate in the composition of 60% HA and 40% β-TCP (particle size between 15-50 nm). Patients in the control group will receive BX (cerabone®, Botiss GmbH, Berlin, Germany). The material is completely anorganic and consists of 100% HA. For this study, the material will be used in granular form (the size of the granules is between 0.5 and 1 mm), mixed with physiological solution prior to placement into the defect.

First surgical phase and healing period Before the procedure, the patient will be administered a 3% chlorhexidine solution to rinse the oral cavity for one minute. Local anesthesia (2% Lidocaine®, Belupo, Koprivnica, Croatia) will be then administered and the surgical field will be covered with sterile drapes. A full-thickness mucoperiosteal flap will be elevated at the extraction site. To perform the tooth extraction atraumatically, the roots of the multirooted teeth will be separated with a drill before extraction. The extraction will be performed with atraumatic instruments, with as little trauma to the alveolus as possible. The alveolus is then carefully examined and curetted to remove granulations and stimulate fresh bleeding in the alveoli. The alveolus will be filled to the edge with I-BCP in the test group and BX in the control group. In the end bone grafting biomaterial is covered with a resorbable native collagen membrane obtained from porcine pericardium (Jason® membrane, Botiss GmbH, Berlin, Germany) in both groups. The mucoperiosteal flap will be then adjusted and closed so that the collagen membrane was completely covered with soft tissue (5.0 monofilament). The patient will be then prescribed an analgesic (400 mg ibuprofen) and instructed to take antibiotics (amoxicillin with clavulanic acid or clindamycin) for the next 7 days. On the 10th day after surgery, the sutures are removed.

A 6-month period of regeneration of the bone defect will follow. Based on the radiographic examination, the selection and positioning of the appropriate implant will be performed.

Second surgical phase Six months after extraction, patients come to the office for placement of a dental implant (Ankylos®, Dentsply Sirona, Charlotte, USA) in the augmented area. The preparation of the patient (rinsing of the oral cavity with an antiseptic solution, local anesthesia, sterile covering of the working area) is the same as for the first surgical procedure. Subsequently, a full-thickness flap is elevated, and a biopsy of the augmented area is taken for histological analysis using a trephine drill (2.5 mm inner diameter; Ustomed® intrumente, Tuttlingen, Germany). It is important to emphasize that the inner diameter of the trephine drill is smaller than that of the final drill used to prepare the implant bed to avoid unnecessary removal of the patient's bone. In addition, each biopsy will be taken from the central part of the augmented area to reduce the possibility of an incorrect biopsy (e.g., bi-opsy of only the native bone that was not augmented with biomaterial).

Histological analysis The trephine drill will be placed in a hermetically sealed plastic tube containing a 4% formaldehyde solution and sent to the histology laboratory for further analysis. The tissue will be fixed in 4% formaldehyde solution for two weeks. Subsequently, the biopsies will be stored in 25% ethylenediaminetetraacetic acid (EDTA) (Decalcifier soft®, Solvagreen®, Karlsruhe, Austria), which is used for gentle decalcification of bone. After decalcification, the tissue will be subjected to a standard protocol in a tissue processor (MTP, SLEE medical GmbH, Mainz, Germany). This will be followed by the formation of paraffin blocks (MPS/P, SLEE medical GmbH, Mainz, Germany). Six consecutive sections of 5 μm thickness will be prepared from each biopsy using a rotary microtome (CUT 4062, SLEE medical GmbH, Mainz, Germany). The specimens will be then stained with Masson trichrome stain and Movat pentachrome stain. Microscopy of the preparations will be performed using a light microscope (Leica DMRB, Leica Microsystems GmbH, Wetzlar, Germany) in conjunction with a video camera (Axio Imager M2, Zeiss, Oberkochen, Germany). Pathohistological analysis will evaluate the tissue response to the implanted biomaterial, i.e., the presence of fibroblasts, blood vessels, neutrophils, monocytes/macrophages, and multinucleated giant cells (MGC).

Histomorphometric processing of the specimens will be performed using the free ImageJ software (https://imagej.nih.gov/ij/download.html). The surface of the new bone, the sur-face of the biomaterial, and the surface of the soft tissue will be marked on the specimens. The surface of the specimen will be then measured, and the following will be calculated from the data obtained: percentage of new bone formed, percentage of biomaterial remaining, and percentage of soft tissue.

Statistical analysis Categorical variables will be reported with absolute and relative frequencies. Differences between categorical variables were tested with the Fisher-Freeman-Halton test.

Normality of distribution will be tested with the Shapiro-Wilk test. Continuous data will be described by the arithmetic mean and standard deviation. Differences in continuous vari-ables will be tested with the Mann-Whitney U test (with corresponding difference and 95% confidence interval of difference).

All P values will be two-sided. The significance level was set at alpha = 0.05. IBM SPSS Statistical software, version 27.0.1, will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years
* patients requires to have at least one tooth predisposed to extraction
* intact physical and mental health
* patient must understand the study protocol
* patient must sign an informed consent.
* the presence of a buccal bone defect such as fenestration or dehiscence.

Exclusion Criteria:

* patients will be excluded from the study if they had at least one of the absolute contraindications to implant prosthetic therapy
* following systemic diseases: uncontrolled diabetes, osteoporosis and osteopenia, and vitamin D deficiency
* bisphosphonate therapy
* glucocorticoid therapy
* hypothyroidism
* uncontrolled cardiovascular disease (hypertension, coronary artery disease, congestive heart failure)
* pregnant or lactating women
* following local factors: use of tobacco products (up to 10 cigarettes per day) and poor oral hygiene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of the newly formed bone, soft tissue and residual biomaterial in bone biopsies harvested 6 months after bone augmentation | Up to 8 months
  Histomorphometric processing of the specimens will be performed using the free ImageJ software (https://imagej.nih.gov/ij/download.html). The surface of the new bone, the surface of the biomaterial, and the surface of the soft tissue will be marked on the specimens. Marked surfaces of the specimen will be then measured, and the following will be calculated from the data obtained: percentage of new bone formed, percentage of biomaterial remaining, and percentage of soft tissue

OTHER OUTCOMES:
Qualitative histological assessment | Up to 8 months
  Tissue response to implanted biomaterial is assessed by descriptive histologic evaluation, i.e., the presence of fibroblasts, blood vessels, neutrophils, monocytes/macrophages, and multinucleated giant cells (MGC).

CONTACTS AND LOCATIONS:
Overall Officials: Marija Candrlic, PhD, Principal Investigator — Faculty of Medicine Osijek
Locations (1):
- Faculty of Medicine Osijek, Osijek, County of Osijek-Baranja, Croatia

IPD SHARING:
Plan to Share IPD: No
I do not plan to make IPD available to other researchers. IPDs will be administrated and stored by one person.

REFERENCES:
- [Background] Candrlic M, Peric Kacarevic Z, Ivanisevic Z, Tomas M, Vcev A, Faj D, Matijevic M. Histological and Radiological Features of a Four-Phase Injectable Synthetic Bone Graft in Guided Bone Regeneration: A Case Report. Int J Environ Res Public Health. 2020 Dec 29;18(1):206. doi: 10.3390/ijerph18010206. PMID 33383971
- [Background] Tomas M, Candrlic M, Juzbasic M, Ivanisevic Z, Matijevic N, Vcev A, Cvijanovic Peloza O, Matijevic M, Peric Kacarevic Z. Synthetic Injectable Biomaterials for Alveolar Bone Regeneration in Animal and Human Studies. Materials (Basel). 2021 May 26;14(11):2858. doi: 10.3390/ma14112858. PMID 34073551